CLINICAL TRIAL: NCT07370636
Title: The Effect of Binaural Beats Stimulation on the Autonomic Nervous System, Considering Kinesiophobia of Reinjuries and Fitness Levels in Professional Athletes With Musculoskeletal Injuries
Brief Title: Binaural Beats Stimulation on the Autonomic Nervous System (ANS), Kinesiophobia and Fitness Levels in Professional Athletes With Musculoskeletal (MSK) Injuries
Acronym: ANS MSK HRV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Collaborators: Attiko Hospital, National and Kapodistrian University of Athens (NKUA) Medical School (Unknown)
Responsible Party: Principal Investigator, Evangelos Kontogiannis, Physiotherapist, PhD candidate, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 62664/07-07-2025
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Kinesiophobia (Fear of Movement); Musculoskeletal Injuries
Keywords: Binaural beats; kinesiophobia; Autonomic nervous system; sympathetic skin response; VO2max; Heart rate variability; grip strength test; pain; anxiety
MeSH Terms: conditions — Kinesiophobia; Pain; Anxiety Disorders | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Binaural beats and guidance (Experimental): The experimental group will participate in a music-based program designed to improve attention, mental alertness, readiness for action and to reduce kinesiophobia. The music track that will be used for this group of participants will include binaural beats and guidance. Participants will receive the music program for 4 weeks / 5 sessions per week, for a total of 20 sessions of 15 minutes each
  Interventions: Device: Auditory stimulation with binaural beats and guidance; Other: Auditory stimulation general characteristics
- No binaural beat but guidance (Placebo Comparator): The Placebo group will participate in a music-based program designed to improve attention, mental alertness, readiness for action and to reduce kinesiophobia. The music track provided to this group will be the same as in the other two groups but it will only include guidance and not binaural beats. Participants will receive the music program for 4 weeks / 5 sessions per week, for a total of 20 sessions of 15 minutes each.
  Interventions: Device: Auditory stimulation without binaural beats; Other: Auditory stimulation general characteristics
- No binaural beat, no guidance (Other): Participants allocated to the control group will undergo a structured music-based intervention designed to enhance attentional focus, mental alertness, and action readiness, while concurrently aiming to reduce kinesiophobia. The music track used for this group will be the same as in the other two groups but it will include neither binaural beats nor guidance. The intervention will be administered for 4 weeks / 5 sessions per week, for a total of 20 sessions of 15 minutes each.
  Interventions: Device: Auditory stimulation with background music; Other: Auditory stimulation general characteristics

INTERVENTIONS:
Device: Auditory stimulation with binaural beats and guidance — The music track will provide auditory stimulation using binaural beats at low beta frequencies (12-15 Hz) accompanied by guided instructions over a low-tempo musical background with a gradual increase in rhythm toward the end of the track.
  Arms: Binaural beats and guidance
Device: Auditory stimulation without binaural beats — The music track will provide auditory stimulation without the use binaural beats (12-15 Hz). It will consist solely of guided instructions delivered over a low-tempo musical background with a gradual increase in rhythm toward the end of the track.
  Arms: No binaural beat but guidance
Device: Auditory stimulation with background music — Auditory stimulation will be delivered exclusively via background music, without the incorporation of binaural beats or guided verbal instructions.
  Arms: No binaural beat, no guidance
Other: Auditory stimulation general characteristics — * Each participant will receive the music track during the pre-training/ pre- competition as a part of the warmup using audible manner
  * All music tracks will employ the same background music, standardized across sessions with identical characteristics, including tempo, frequency, and other acoustic parameters, to ensure consistency throughout the intervention.
  * Questionnaires are going to be used to evaluate kinesiophobia, sport anxiety, competitions and pain beliefs and perceptions pre and post the music intervention for all participants.

SUMMARY:
The purpose of the current study is to investigate the effectiveness of binaural beat stimulation on the autonomic nervous system (ANS), taking into account kinesiophobia related to reinjury and fitness levels in professional athletes with musculoskeletal injuries. The study hypothesis is that binaural beats will have beneficial effects by reducing ANS activity, primarily through modulation of parasympathetic nervous system (PNS) activity, as well as by reducing kinesiophobia related to reinjury and enhancing fitness levels in this population.

Researchers will compare binaural beat stimulation to a placebo condition and to a condition without binaural beats in order to evaluate and compare the effects of those three conditions on psychological and physiological parameters in professional athletes with musculoskeletal injuries.

Participants will:

* Receive receive music intervention either with binaural beat stimulation or placebo or music without binaural beats before their training sessions and competitions for a period of four weeks.
* Maintain a diary to document each session of the music-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Professional athletes in open-skill sports
* Age 18-25 years old
* Participation in national and/or international professional championships for ≥ 5 years
* Athletes with previous lower limb musculoskeletal injuries within the past three months or longer
* Athletes with previous lower limb musculoskeletal injuries who have been fully rehabilitated.
* Injuries sustained during any training period or competitive event
* Provoke injuries during any training period or competitive event
* Athletes with Kinesiophobia who have presented Tampa of Scale Kinesiophobia (TSK) questionnaire scores ranging from 17 to 37
* Athletes with Anxiety who have presented Sport Competition Anxiety Test (SCAT) questionnaire scores more than 17
* Frequency of engaging in sports 3-5 times per week (training, competitions)
* Duration of each training session not exceeding 90 minutes
* Athletes with adequate proficiency in the English language

Exclusion Criteria:

* Amateur and recreational athletes in open-skill activities
* Athletes ≤ 17 and ≥ 26 years old
* Athletes in close-skill sports
* Athletes with current musculoskeletal injuries (< 3 months)
* Athletes with poor rehabilitation of sport injuries
* Athletes with musculoskeletal injuries of upper limbs and trunk
* Athletes with musculoskeletal injuries during off-season periods
* Athletes with recent surgery
* Athletes with a concussion that occurred during training or competition
* Athletes with psychological and neurological problems
* Athletes with hearing impairment
* Athletes with inadequate proficiency in the English language

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Sympathetic Skin Response | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks
  Sympathetic Skin Response (SSR) test will be used to assess the changes of the Autonomic Nervous System (ANS). SSR will be assessed by calculating the latency and the amplitude. The Latency was measured from the onset of the stimulus artefact to the first deflection from baseline (in seconds) and amplitude was measured peak-to-peak (from negative to positive peak, in millivolts). The Sympathetic Skin Response will be carried out using Electromyography (EMG). Electrical stimuli were delivered to the right wrist at an intensity of 75 mA and a duration of 0.1 ms. The band-pass filter was set between 0.5 and 2000 Hz. Five stimuli were administered unpredictably at random intervals of at least 30 seconds. The shortest latency and the highest amplitude response values among the five responses were used for statistical analysis. Parameters included in the analysis were: SSR upper limb latency, SSR upper limb amplitude, SSR lower limb latency, and SSR lower limb amplitude.
Tampa Scale of Kinesiophobia (TSK-17) | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks
  Tampa Scale of Kinesiophobia questionnaire (TSK-17) will be used translated to Greek. It has been tested for its reliability and validity. Scale from 17 to 68. 17 means the person experiences low level of kinesiophobia and 68 means the person experiences high level of kinesiophobia.
Aerobic capacity | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  An incremental exercise test will be used to assess the aerobic capacity. This method is commonly used to evaluate maximal oxygen uptake (VO₂max) and involves a protocol of progressively increasing exercise intensity until volitional exhaustion. Participants will run on a motorized treadmill set at a constant incline of 0%. Running speed will begin at approximately 8-9 km/h and will increase by 1 km/h at the end of each 1-minute stage. Respiratory variables will be continuously measured on a breath-by-breath basis using a gas analysis system. The test will be terminated when participants reach volitional exhaustion, when oxygen uptake values plateau or decrease despite further increases in workload and ventilation or when the respiratory exchange ratio exceeds 1.10. Total test duration is expected to be approximately 8-12 minutes.
Heart Rate Variability (HRV) | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  Heart Rate Variability (HRV) is a tool to assess the Autonomic Nervous System function. HRV will be recorded using a telemetric heart rate monitor (Polar H10). Recordings will be conducted in a quiet, calm room, with participants in the supine position. Participants will be instructed not to move, talk, and to breathe normally while remaining supine during the recording. All participants will perform an incremental exercise test on a treadmill at a constant 0% incline, with intensity gradually increasing every minute. Prior to the test, participants will lie supine for 5 minutes while resting HRV is recorded. Participants will then follow the exercise protocol and at the end of the exercise, they will be asked to remain supine for 15 minutes. The time required for HRV to return to each participant's resting level will be recorded. The test will be automatically terminated once participants reach 85% of their maximum heart rate (HRmax) or voluntarily.

SECONDARY OUTCOMES:
Sport competition anxiety | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  Sport competition anxiety questionnaire (SCAT) will be used translated to Greek. It has been tested for its reliability and validity. Scale from 10 to 30. Scores under 17 show low level of competition anxiety. Scores over 24 show high level of competition anxiety.
Pain Beliefs and Perceptions Inventory | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  Pain Beliefs and Perceptions Inventory questionnaire (PBPI-16) will be used translated to Greek. It has been tested for its reliability and validity. Scale from -32 to 32. -32 means the person does not express negative beliefs, 32 means the person expresses negative beliefs.
Hand Grip Strength Test | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  The Hand Grip Strength Test will be used to assess grip strength through the performance of a maximal voluntary contraction. A portable Kinvent hand dynamometer will be used for the assessment. The test will be performed in a seated position with the shoulder in a neutral position, the elbow flexed at 90° without support, the forearm in a neutral position, and the wrist positioned between 0° and 30° of dorsiflexion and 0°-15° of ulnar deviation. Participants will perform three maximal efforts, each lasting 30 seconds, with a 1-minute rest period between attempts. The test will be conducted in the same manner for both upper limbs. For statistical analysis, the mean value of the three trials will be calculated separately for each upper limb.
Blood lactate concentration | Changes from baseline up to 4 weeks; changes from baseline up to 8 weeks.
  Blood lactate concentration will be measured before the incremental exercise test and at the end of the test.

REFERENCES:
- [Background] Ingendoh RM, Posny ES, Heine A. Binaural beats to entrain the brain? A systematic review of the effects of binaural beat stimulation on brain oscillatory activity, and the implications for psychological research and intervention. PLoS One. 2023 May 19;18(5):e0286023. doi: 10.1371/journal.pone.0286023. eCollection 2023. PMID 37205669
- [Background] Delleli S, Ouergui I, Ballmann CG, Messaoudi H, Trabelsi K, Ardigo LP, Chtourou H. The effects of pre-task music on exercise performance and associated psycho-physiological responses: a systematic review with multilevel meta-analysis of controlled studies. Front Psychol. 2023 Nov 23;14:1293783. doi: 10.3389/fpsyg.2023.1293783. eCollection 2023. PMID 38078229
- [Background] Cici R, Bulbuloglu S, Kapikiran G. Effect of meditation music and comedy movie interventions on postoperative kinesiophobia and pain in patients undergoing total knee arthroplasty. ANZ J Surg. 2023 Jan;93(1-2):302-309. doi: 10.1111/ans.18209. Epub 2022 Dec 14. PMID 36515211
- [Background] Chee ZJ, Chang CYM, Cheong JY, Malek FHBA, Hussain S, de Vries M, Bellato A. The effects of music and auditory stimulation on autonomic arousal, cognition and attention: A systematic review. Int J Psychophysiol. 2024 May;199:112328. doi: 10.1016/j.ijpsycho.2024.112328. Epub 2024 Mar 6. PMID 38458383
- [Background] Ballmann CG. The Influence of Music Preference on Exercise Responses and Performance: A Review. J Funct Morphol Kinesiol. 2021 Apr 8;6(2):33. doi: 10.3390/jfmk6020033. PMID 33917781
- [Background] Bordeleau M, Vincenot M, Lefevre S, Duport A, Seggio L, Breton T, Lelard T, Serra E, Roussel N, Neves JFD, Leonard G. Treatments for kinesiophobia in people with chronic pain: A scoping review. Front Behav Neurosci. 2022 Sep 20;16:933483. doi: 10.3389/fnbeh.2022.933483. eCollection 2022. PMID 36204486
- [Background] Wahbeh H, Calabrese C, Zwickey H. Binaural beat technology in humans: a pilot study to assess psychologic and physiologic effects. J Altern Complement Med. 2007 Jan-Feb;13(1):25-32. doi: 10.1089/acm.2006.6196. PMID 17309374
- [Background] Ambegaonkar JP, Jordan M, Wiese KR, Caswell SV. Kinesiophobia in Injured Athletes: A Systematic Review. J Funct Morphol Kinesiol. 2024 Apr 19;9(2):78. doi: 10.3390/jfmk9020078. PMID 38651436
- [Background] Franco-Alvarenga, P., Brietzke, C., Canestri, R., & Pires, F. (2019). Psychological responses of music on physical performance: A critical review. Revista Brasileira de Ciência e Movimento, 2019;27(2):218-224.
- [Background] Fukumoto Y, Tsuji Y, Kakuda A, Hori R, Kitano M, Sakamoto K, Kudo S. Evaluation of autonomic nervous system responses during isometric handgrip exercise using nonlinear analysis of heart rate variability. J Phys Ther Sci. 2022 Oct;34(10):689-693. doi: 10.1589/jpts.34.689. Epub 2022 Oct 1. PMID 36213191